CLINICAL TRIAL: NCT00810719
Title: Phase II Study of Gemcitabine and Intermittent Erlotinib in Advanced Pancreatic Cancer
Brief Title: Gemcitabine and Erlotinib in Treating Patients With Metastatic or Recurrent Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#211; 232494 (Other: UC Davis); OSI 4132s (Other: Genentech); P30CA093373 (NIH)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and Erlotinib (Experimental): The dose for gemcitabine is 1,000 mg/m2 administered over 30 minutes as an intravenous infusion. The doses are administered weekly for 3 weeks (Days 1, 8 and 15) followed by one week of rest during which gemcitabine is not given. This 4 week period (28 days) constitutes a cycle.Erlotinib will be dosed at 150mg orally (tablets) on days 2-5, 9-12, and 16-26 of a 28 day cycle.
  Interventions: Drug: Erlotinib; Drug: gemcitabine

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be administered at 150 mg once daily by mouth on the following schedule: days 2-5, 9-12,16-26.
  Other Names: Tarceva
Drug: gemcitabine — The dose for gemcitabine is 1,000 mg/m2 administered over 30 minutes as an intravenous infusion. The doses are administered weekly for 3 weeks (Days 1, 8 and 15) followed by one week of rest during which gemcitabine is not given. This 4 week period (28 days) constitutes a cycle.
  Other Names: Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with erlotinib works in treating patients with metastatic or recurrent pancreatic cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study.

Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15 and oral erlotinib hydrochloride on days 2-5, 9-12, and 16-26. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Archived tumor tissue samples are analyzed for the expression of EGFR, HER3, HER2, downstream signaling molecules, and other molecular markers by immunohistochemistry and RT-PCR. The presence of aberrant gene copy numbers (amplification and polysomy) for EGFR, HER3, and HER2 are determined by FISH. Blood samples are collected at baseline and periodically during study for polymorphism analysis and correlative molecular analysis of surrogate endpoint biomarkers.

After completion of study therapy, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced, metastatic or recurrent pancreatic carcinoma
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension
* No prior chemotherapy for metastatic or recurrent disease is allowed. Prior adjuvant chemotherapy is allowed provided that patients did not receive gemcitabine and the chemotherapy was completed > six months prior to initiation of study therapy. Prior erlotinib therapy is not allowed
* Available tumor specimen that was obtained at the time of diagnosis and/or prior to study entry is highly encouraged
* Age ≥ 18 years
* Life expectancy greater than 3 months
* Zubrod performance status ≤ 2
* Patients must have normal organ and marrow function as defined below:
* leukocytes ≥ 3,000/μL
* absolute neutrophil count ≥ 1,500/ μL
* platelets ≥ 100,000/ μL
* total bilirubin ≤ 1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) ≤ 3 X institutional upper limit of normal, unless the liver is involved with tumor, in which case the AST/ALT must be ≤ 5 X institutional upper limit of normal
* creatinine clearance ≥ 50 mL/min/1.73 m2, as measured by 24hour collection OR
* creatinine ≤ 1.5 X institutional upper limit of normal
* The effects of erlotinib and gemcitabine on the developing human fetus at the recommended therapeutic doses are unknown. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib or gemcitabine.
* Secondary primary malignancy. Concurrent or history of another malignancy < 5 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because erlotinib and gemcitabine have the potential for teratogenic or abortifacient effects. Breastfeeding should be discontinued if the mother is treated with study drugs.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California

REFERENCES:
- [Result] Semrad T, Barzi A, Lenz HJ, Hutchins IM, Kim EJ, Gong IY, Tanaka M, Beckett L, Holland W, Burich RA, Snyder-Solis L, Mack P, Lara PN Jr. Pharmacodynamic separation of gemcitabine and erlotinib in locally advanced or metastatic pancreatic cancer: therapeutic and biomarker results. Int J Clin Oncol. 2015 Jun;20(3):518-24. doi: 10.1007/s10147-014-0730-2. Epub 2014 Aug 5. PMID 25091263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at University of California Davis and the University of Southern California.
Period: Overall Study
Arm/Group | Gemcitabine and Erlotinib
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Erlotinib
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Defined as the time from first day of treatment to the first observation of disease progression or death due to any cause. If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Erlotinib
Number analyzed (Participants) | 30
months | 2.07 [1.87 to 5.50]

2. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Population: Two patients withdrew consent in the first cycle and were not evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine and Erlotinib
Number analyzed (Participants) | 28
percentage of participants | 11

3. Secondary Outcome: Overall Survival
Description: Overall survival will be followed for survival every three months until documented progression, death or study termination. If a participant is still alive, survival time is censored at the time of last follow-up.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Erlotinib
Number analyzed (Participants) | 30
months | 5.67 [2.83 to 11.87]

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: Start of study treatment and ends 30 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier.
Arm/Group | Gemcitabine and Erlotinib
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Erlotinib (N=30)
Lung Infection (Infections and infestations) | 1
Fatigue (General disorders) | 2
Mental Status Changes (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Skin Infection (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Erlotinib (N=30)
Hemoglobin (Blood and lymphatic system disorders) | 17
Leukopenia (Blood and lymphatic system disorders) | 13
Lymphopenia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Fatigue (General disorders) | 8
Weight Loss (General disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 16
Anorexia (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 9
Mucositis (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 9
Taste Alteration (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Alkaline Phosphatase (Metabolism and nutrition disorders) | 8
ALT (Metabolism and nutrition disorders) | 8
AST (Metabolism and nutrition disorders) | 8
Hyperbilirubinemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Due to funding considerations, the study was closed after thirty participants were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No